CLINICAL TRIAL: NCT00530270
Title: Randomized Trial of Oral Dexamethasone for Acute Chest Syndrome
Brief Title: Dexamethasone to Treat Acute Chest Syndrome in People With Sickle Cell Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was closed June 23, 2008 due to low enrollment.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr. Charles Quinn, Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 516; U54HL070587 (NIH); U54HL070587-07 (NIH)
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Results first posted 2009-12-31 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-03

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell Disease; ACS; Acute Chest Syndrome; Hgb SS; Hgb Sβ0; Dexamethasone
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Individuals meeting entry criteria will be randomized to receive dexamethasone 0.3 mg/kg (12 mg maximum single dose). The study drug will be given by mouth every 12 hours until discharge from the hospital or for a maximum of 4 doses (2 days), whichever occurs first. Thereafter, study drug will be tapered over 6 days for a total duration of therapy not to exceed 8 days.
  Arms: Dexamethasone
Drug: Placebo — Individuals meeting entry criteria will be randomized to receive 0.3 mg/kg (12 mg maximum single dose) of placebo. The study drug will be given by mouth every 12 hours until discharge from the hospital or for a maximum of 4 doses (2 days), whichever occurs first. Thereafter, study drug will be tapered over 6 days for a total duration of therapy not to exceed 8 days.
  Arms: Placebo

SUMMARY:
People with sickle cell disease (SCD) may develop acute chest syndrome (ACS), which is a common and serious lung condition that usually requires hospitalization. Dexamethasone is a medication that may decrease hospitalization time for people with ACS, but it may also bring about new sickle cell pain. This study will evaluate the effectiveness of a dexamethasone regimen that includes a gradual dose reduction at decreasing hospitalization and recovery time in people with SCD and ACS.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder. Symptoms include anemia, infections, organ damage, and intense episodes of pain, which are called "sickle cell crises." ACS is a life-threatening, lung-related complication of SCD that can lower the level of oxygen in the blood. Repeat occurrences of ACS can cause lung damage. It is the second most common cause of hospitalizations among people with SCD and accounts for more than 25% of premature deaths in people with SCD. Symptoms of ACS include fever, chest pain, cough, and breathing difficulties. ACS can appear suddenly and often requires immediate hospitalization and treatment, including antibiotics, supplemental oxygen, and blood transfusions. Previous studies have shown that dexamethasone, a type of steroid medication that blocks inflammation, can decrease hospitalization time for people with ACS; however, some participants in these earlier studies were re-hospitalized due to new sickle cell pain. Slowly decreasing the dosage of dexamethasone over a period of time may decrease the chance that new sickle cell pain will occur. The purpose of this study is to evaluate the effectiveness of a dexamethasone regimen that includes a gradual dose reduction at decreasing hospitalization and recovery time in people with SCD and ACS.

This study will enroll people with SCD who are hospitalized and have been diagnosed with ACS within the past 24 hours. Participants will be randomly assigned to receive either dexamethasone or placebo on a daily basis for 8 days. Every 2 days the medication dose will be gradually reduced. While in the hospital, participants will receive usual care for ACS, including antibiotics, pain control medication, intravenous fluids, and other needed treatments. Each day, participants will undergo a physical exam, a pain assessment score, a test to measure the oxygen level in the body, blood collection, and, if needed, a chest x-ray. Vital signs and blood pressure measurements will be taken every 4 hours. Study staff will document the amount of pain medication, blood transfusions, oxygen, and breathing treatments participants receive.

Upon leaving the hospital, follow-up visits will occur 1 week after participants were originally admitted to the hospital (participants who are still hospitalized at this time will not attend this visit) and 1 month after hospital discharge. At both visits, information on hospital visits for pain treatment and blood transfusions will be collected, and evaluations performed earlier in the study will be repeated. The second visit will also include lung function tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell anemia (Hgb SS) or sickle-β0-thalassemia (Hgb Sβ0)
* Current episode of ACS, defined as a new lobar or segmental pulmonary infiltrate seen on a chest radiograph and two or more of the following findings:

  1. Temperature of 38.5°C or higher
  2. Tachypnea (i.e., rapid breathing)
  3. Dyspnea or increased work of breathing
  4. Chest wall pain
  5. Oxygen saturation of less than 90% in room air by pulse oximetry
* Current episode of ACS diagnosed in the 24 hours prior to study entry
* Ability to take medication in capsule form

Exclusion Criteria:

* Prior participation in this study
* Diagnosed with any medical condition that will likely be worsened by corticosteroid therapy, including any of the following conditions:

  1. Diabetes mellitus
  2. High blood pressure
  3. Esophageal or gastrointestinal ulceration or bleeding
  4. Known avascular necrosis
* Diagnosis of ACS in the 6 months prior to study entry
* Treatment with oral or parenteral corticosteroid therapy for any reason in the 14 days prior to study entry
* Use of inhaled corticosteroids or systemic corticosteroids for respiratory illness in the 3 months prior to study entry
* Long-term lung condition that requires treatment with corticosteroids
* Participation in a program of chronic transfusions that ended fewer than 4 months ago. A program of chronic transfusions includes a regimen of serial simple or exchange transfusions given at least every 6 weeks for at least three consecutive transfusions for the prevention of SCD-related complications.
* Pregnant
* Treatment with any investigational drug in the 90 days prior to study entry
* History of either tuberculosis or a positive skin test for tuberculosis
* Known HIV infection or a current systemic fungal infection

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Quinn, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (6):
- United States (6):
  - University of California - Davis, Sacramento, California
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital Boston, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - St. Christopher's Hospital, Philadelphia, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas

REFERENCES:
- [Derived] Quinn CT, Stuart MJ, Kesler K, Ataga KI, Wang WC, Styles L, Smith-Whitley K, Wun T, Raj A, Hsu LL, Krishnan S, Kuypers FA, Setty Y, Rhee S, Key NS, Buchanan GR; Investigators of the Comprehensive Sickle Cell Centers. Tapered oral dexamethasone for the acute chest syndrome of sickle cell disease. Br J Haematol. 2011 Oct;155(2):263-7. doi: 10.1111/j.1365-2141.2011.08827.x. Epub 2011 Aug 16. PMID 21848879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from October 2006 through June 2008 at 10 sites across the United States. Due to the acute nature of the disease under study, subjects were recruited in a hospital, frequently in the Emergency Department.
Pre-assignment Details: No events excluded patients following enrollment, but prior to group assignment. Group assignments were made at enrollment.
Groups:
- Dexamethasone; Placebo: 0.3 mg/kg (12 mg maximum single dose) every 12 hours until discharge from the hospital or for a maximum of 4 doses, whichever comes first. Thereafter, study drug will be tapered over 6 days (not to exceed 8 days).
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 18.8 (14.08) | 15.8 (12.81) | 17.3 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Log (Natural) of Duration of Signs and Symptoms of Acute Chest Syndrome (ACS) or Duration of Hospitalization, Whichever is Less
Description: Resolution of symptoms of ACS includes respiratory rate <= upper limit of normal +2, no work of breathing (retractions, nasal flaring, and use of accessory muscles), thoracic pain <= 4, no use of supplemental oxygen, no use of ventilary support, and saturation of peripheral oxygen (Sp02) >= steady state value -2. Symptoms were measured every 4 hours from the first dose of study drug to resolution of symptoms or hospital discharge.
Time Frame: Measured from first dose to end of the hospital stay, no maximum number of days
Population: Subject without major protocol violation and received treatment.
Measure: Log Mean (Standard Deviation); unit: hours (log transformed)
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 5 | 6
hours (log transformed) | 2.4 (1.23) | 3.5 (0.60)
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; The null hypothesis of no difference in the log duration of signs and symptoms or hospitalization between the two treatment groups was tested using an F test from a generalized mixed model with fixed effects for treatment group, age group and ACS severity. Please note that the study was stopped prematurely so only 11 of the 112 originally planned were included in the analysis; Test type: Superiority or Other; p = 0.127, Mixed Models Analysis — A two-sided alpha of 0.05 was used. No multiple comparison adjustments were made

2. Secondary Outcome: Rating of Pain
Description: Change from baseline rating of pain from randomization (baseline) to discharge from the hospital, evaluated every 4 hours. Pain was rated on the Oucher Scale for the pediatric population or numeric rating scale for the adult population, both 0 to 10 with 0 indicating no pain and 10 indicating severe pain.
Time Frame: Measured at the end of the hospital stay
Population: Subject without major protocol violation and received treatment.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 5 | 6
Units on a scale
  Thoracic | -3.8 (1.34) | -4.1 (1.26)
  Non-thoracic | -2.0 (1.35) | -1.4 (1.28)
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.801, Mixed Models Analysis — A two-sided alpha of 0.05 was used. No multiple comparison adjustments were made

3. Secondary Outcome: Duration of Hospitalization
Description: Duration in hours from treatment start time to hospital discharge.
Time Frame: Measured at the end of hospital stay, no maximum number of days
Population: Subject without major protocol violation and received treatment.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 5 | 6
Hours | 41.5 (9.03) | 62.3 (14.27)
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis — A two-sided alpha of 0.05 was used. No multiple comparison adjustments were made; Different error variance estimates were allowed for the two treatment groups

4. Secondary Outcome: Duration of Supplemental Oxygen
Description: Time period between the supplemental oxygen start date/time and first dose date/time, whichever is later, and the supplemental oxygen stop date/time
Time Frame: Measured at the end of hospital stay
Population: Subject without major protocol violation and received treatment.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 5 | 6
Hours | 17.5 (0) | 41.2 (22.22)
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.876, Mixed Models Analysis — A two-sided alpha of 0.05 was used. No multiple comparison adjustments were made; Different error variance estimates were allowed for the two treatment groups

5. Secondary Outcome: Duration of Hypoxemia (Low Blood Oxygen)
Description: Sum of time periods when subject was hypoxemic (Sp02 value less than 92%) since the first dose date/time
Time Frame: Measured at the end of hospital stay
Population: Subject without major protocol violation and received treatment.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 5 | 6
Hours | 13.8 (0) | 38.4 (22.18)
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.770, Mixed Models Analysis — A two-sided alpha of 0.05 was used. No multiple comparison adjustments were made; Different error variance estimates were allowed for the two treatment groups

ADVERSE EVENTS:
Arm/Group | Dexamethasone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=6) | Placebo (N=6)
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=6) | Placebo (N=6)
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Primary limitation of this study is that is was terminated prior to enrolling all of the subjects necessary to address the primary question.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No